CLINICAL TRIAL: NCT02609243
Title: Diabetes Nutrition Algorithm - Prediabetes (Dietary Strategies in the Prevention of Diabetes Mellitus Type 2 in a High-risk Cohort)
Brief Title: Diabetes Nutrition Algorithm - Prediabetes
Acronym: DiNA-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Diabetes Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, Director / Department for Clinical Nutrition, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DiNA-P
Record Dates: First submitted 2015-03-23; First posted 2015-11-20 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Prediabetes; Diabetes Mellitus Type 2; Obesity; NAFLD; Dyslipoproteinemia
Keywords: prediabetes; diabetes mellitus type 2; obesity; NAFLD; dyslipoproteinemia
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Obesity; Non-alcoholic Fatty Liver Disease; Dyslipidemias | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- intensive consulting, conventional diet (Active Comparator): subjects receive 16 units of nutritional consulting, first 3 weeks of intervention phase are designed as a conventional hypocaloric low-fat diet referring to DGE guidelines (below 30 % fat), followed by 11 months of isocaloric-to-moderate-hypocaloric low-fat diet (below 30 kcal% fat ) - dietary intervention without supplement
  Interventions: Behavioral: dietary consulting
- conventional consulting, low-carb diet (Active Comparator): subjects receive 8 units of nutritional consulting, first 3 weeks of intervention phase are designed as a very-low calory ketogenic (low-carb) diet (< 40 g CH / day), following 11 months are restricted to not more than 40 % energy intake by carbohydrates under isocaloric-to-moderate-hypocaloric conditions - dietary intervention without supplement
  Interventions: Behavioral: dietary consulting
- conventional consulting, conventional diet (Active Comparator): subjects receive 8 units of nutritional consulting, first 3 weeks of intervention phase are designed as a conventional hypocaloric low-fat diet referring to DGE guidelines (below 30 % fat), followed by 11 months of isocaloric-to-moderate-hypocaloric low-fat diet (below 30 kcal% fat) - dietary intervention without supplement
  Interventions: Behavioral: dietary consulting
- intensive consulting, low-carb diet (Active Comparator): subjects receive 16 units of nutritional consulting, first 3 weeks of intervention phase are designed as a very-low calory ketogenic (low-carb) diet (< 40 g CH / day), following 11 months are restricted to not more than 40 % energy intake by carbohydrates under isocaloric-to-moderate-hypocaloric conditions - dietary intervention without supplement
  Interventions: Behavioral: dietary consulting

INTERVENTIONS:
Behavioral: dietary consulting — dietary consulting implies specific dietary advice based on pre-interventional self-report regarding food intake; consulting focuses on nutrient content, calory intake, weight loss; with regard to randomisation consulting intensity and content varies
  Other Names: dietary intervention without supplement

SUMMARY:
Prediabetes, defined by either impaired fasting glucose and/or impaired glucose tolerance, is a known high-risk condition predisposing to future diabetes mellitus type 2. Strategies to prevent progression from prediabetes to diabetes have been widely studied, however, without striking long-term effects of any kind of intervention (pharmacological, behavioral...). The investigators therefore investigate certain nutritional approaches concerning nutrient content and favorable food components, targeting metabolic improvement.

DETAILED DESCRIPTION:
Prediabetes, defined by either impaired fasting glucose and/or impaired glucose tolerance, is a known high-risk condition predisposing to future diabetes mellitus type 2. Strategies to prevent progression from prediabetes to diabetes have been widely studied, however, without striking long-term effects of any kind of intervention (pharmacological, behavioral...). The investigators therefore investigate certain nutritional approaches concerning nutrient content and favorable food components, targeting metabolic improvement.

The main comparison will assess differences in metabolic outcome due to low-carb or low-fat dietary intervention in short- and long-term design.

Additionally, the role of PUFA will be assessed during long-term intervention to achieve better maintenance of metabolic improvements from the first study phase.

ELIGIBILITY:
Inclusion Criteria:

* impaired fasting glucose (IFG) fasting blood glucose 100-126 mg/dl

and/or

* impaired glucose tolerance (IGT) 75 g OGTT 120 minutes: 140-200 mg/dl

Exclusion Criteria:

* current pregnancy or breastfeeding
* BMI > 45 kg/m²
* Diabetes mellitus Typ 1 or 2
* serious disease e.g symptomatic coronary heart disease
* serious symptomatic malignant disease (weight loss > 10% within the last 6 month)
* severe liver or kidney disease ( an increase in transaminases > 3 times than the upper limit of the standardized range, GFR < 50 ml/min/1,73m²)
* systemic infection (CRP > 1 mg/dl)
* severe mental illness
* drug abuse
* treatment with steroids
* potentially incompliant subjects
* exclusion criteria for magnetic resonance tomography
* any kind of metal in or on the body: cardiac pacemakers prosthetic heart valves metal prosthesis magnetic implanted metallic parts contraceptive coil metal fragments/ grenade shrapnel fixed braces acupuncture needles insulin pump intraport etc. Field strength > 3 Tesla further tattoos, permanent make-up
* persons with limited thermosensory or heightened sensitivity to heating
* persons where cardiovascular disease cannot be ruled out by examination
* persons with heightened sensitivity to loud noise or diseases of the ear
* used closed whole body scanner: claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
change in postprandial glycaemia (2h plasma glucose level of the 75 g oral glucose tolerance test (OGTT)) | 3 weeks, 6 months, 1 year, 3 years
change in hepatic fat content confirmed by proton magnetic resonance spectroscopy by 3 T MR imaging | 3 weeks, 6 months, 1 year, 3 years

SECONDARY OUTCOMES:
change in insulin sensitivity confirmed by 75 g oral glucose tolerance test (OGTT) | 3 weeks, 6 months, 1 year, 3 years
  insulin resistance is calculated as follows:
  Insulinogenic index (IGI) = (I30 - I0) / (G30 - G0) ISIest= 10000/²√ ((G0 x I0) x ((G0+G30+G60+G90+G120)/5) x ((I0+I30+I60+I90+I120)/5))
change in insulin secretion confirmed by 75 g oral glucose tolerance test (OGTT) | 3 weeks, 6 months, 1 year, 3 years
  insulin resistance is calculated as follows:
  Insulinogenic index (IGI) = (I30 - I0) / (G30 - G0) ISIest= 10000/²√ ((G0 x I0) x ((G0+G30+G60+G90+G120)/5) x ((I0+I30+I60+I90+I120)/5))
change in distribution of body fat confirmed by MR-Imaging by 3 T whole body imager | 3 weeks, 6 months, 1 year, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof. Dr., Principal Investigator — German Institute of Human Nutrition
Locations (2):
- Germany (2):
  - German Institut for Human Nutrition; Department for Clinical Nutrition, Bergholz-Rehbrücke, Brandenburg
  - German Institute for Human Nutrition, Department for Clinical Nutrition, Berlin